CLINICAL TRIAL: NCT04165759
Title: Preoperative Evaluation of High-resolution Computed Tomography to Predict Pathologic Tumor Invasion in Ground-glass Opacity Featured Lung Adenocarcinoma
Brief Title: HRCT in Prediction of Tumor Invasion in GGO Lung Adenocarcinoma (ECTOP-1008)
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Collaborators: Fujian Medical University Union Hospital (Other); Shandong First Medical University Affiliated Liaocheng Second Hospital (Unknown); Jiangdu People's Hospital, Yangzhou (Unknown)
Responsible Party: Principal Investigator, Haiquan Chen, Director of Department of thoracic surgery and multidisciplinary group of thoracic oncology, Fudan University
Other Study IDs: PRSHRCT
Record Dates: First submitted 2019-11-14; First posted 2019-11-18 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Adenocarcinoma of Lung
MeSH Terms: conditions — Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Lung surgical specimens
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients: Patients with lung cancer who are candidates for surgery.

SUMMARY:
This study is one of Eastern Cooperative Thoracic Oncology Projects (ECTOP-1008). It aims to evaluate the correlation between radiological diagnosis based on HRCT and pathological invasiveness.Investigators observe the radiological features and the correlation with the postoperative pathological findings.

DETAILED DESCRIPTION:
Preoperative evaluation of pathologic tumor invasion of ground glass opacity (GGO) featured lung adenocarcinoma is important for selection of appropriate surgical extent. Whether thoracic high-resolution computed tomography (HRCT) scan could precisely predict pathologic tumor invasion remains unknown. Patients with peripheral GGO nodules (GGNs) would be enrolled, and HRCT with target scan would be performed preoperatively. Pathologic tumor invasion (invasive adenocarcinoma [IAD] versus adenocarcinoma in situ [AIS]/minimally invasive adenocarcinoma [MIA]) would be evaluated according to radiologic parameters of HRCT before surgery. Primary endpoint of this trial is the diagnostic sensitivity of pathologic tumor invasion evaluated by HRCT. Secondary endpoint is the diagnostic value of radiologic parameters of HRCT for pathologic tumor invasion of GGO featured lung adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

(1) GGNs on HRCT scan; (2) clinical stage IA; (3) simultaneously no more than three nodules; (5) Age ranging from 15 to 85 years.

Exclusion Criteria:

(1) pathologically confirmed non-adenocarcinoma; (2) patients who did not receive surgery.

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: East Asian population
Sampling Method: Probability Sample
Enrollment: 620 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity | Pathologic reports were available, usually 1 month after surgery
  Diagnostic sensitivity of pathologic tumor invasion evaluated by HRCT

SECONDARY OUTCOMES:
Value of radiologic parameters for tumor invasion | Pathologic reports were available, usually 1 month after surgery
  The receiver operating characteristic curve (ROC curve) and the area under the ROC curve (AUC) of the invasion prediction model based on radiologic parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Haiquan Chen, Principal Investigator — Fudan University
Locations (2):
- China (2):
  - Fudan University Cancer Center, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
The IPD could be shared if a reasonable request was proposed.
Supporting Information: Study Protocol, ICF
Time Frame: The IPD could be shared if a reasonable request was proposed.
Access Criteria: An individual researcher could sent a mail to hqchen1@yahoo.com for these data.